CLINICAL TRIAL: NCT05555745
Title: Audio-based Mental Health Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Michelle G. Newman, Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020667
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Depressive Symptoms
Keywords: digital interventions; mhealth; depression; behavioral activation; podcasts; self-help
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Audio-based behavioral activation intervention (Experimental): This intervention consists of two audio-based sessions delivered one week apart. The first session lasts approximately 30 minutes, and the second session lasts approximately 15 minutes. The sessions are audio recordings. The first session introduces behavioral activation and provides instruction for how to schedule and engage in positively reinforcing activities. The second session recaps the principles of behavioral activation and guides participants through methods of troubleshooting. After each session, participants are asked to create an activity schedule for the coming week. Then, each day in the week following each session, participants receive an email with a survey asking them to report on their activity and mood in the previous day.
  Interventions: Device: Audio-based behavioral activation intervention
- Audio-based self-monitoring intervention (Active Comparator): This intervention consists of two audio-based sessions delivered one week apart. The first session lasts approximately 30 minutes, and the second session lasts approximately 15 minutes. The sessions are audio recordings. The first session introduces information about emotion and provides instruction for how to track emotion using self-monitoring. The second session provides more information about emotion and recaps instructions for self-monitoring. Each day in the week following each session, participants receive an email with a survey asking them to report on their mood in the previous day.
  Interventions: Device: Audio-based self-monitoring intervention

INTERVENTIONS:
Device: Audio-based behavioral activation intervention — Access to audio-based behavioral activation intervention
  Arms: Audio-based behavioral activation intervention
Device: Audio-based self-monitoring intervention — Access to audio-based self-monitoring intervention
  Arms: Audio-based self-monitoring intervention

SUMMARY:
This is a study on an audio-based digital intervention designed to reduce symptoms of depression. Participants who experience at least moderate symptoms of depression will be invited to participate in the study. Participants will be randomly assigned to receive one of two audio-based digital interventions. The experimental intervention based on behavioral activation treatment for depression. The control intervention is based on self-monitoring. Depression symptoms and related mental health symptoms, as well as experiences with the intervention, will be assessed at baseline (pre-randomization), mid-intervention (1 week post-randomization), post-intervention (2 weeks post-randomization) and follow-up (5 weeks post-randomization)

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 or older
* Score in the moderate or higher range on the BDI-FastScreen
* Moderate or higher depression confirmed by DIAMOND interview
* Proficient English reading, writing, and speaking ability
* Able to provide consent
* Provide informed consent

Exclusion Criteria:

* Below 18 years of age
* Score below the moderate range on the BDI-FastScreen
* DIAMOND interview does not confirm moderate or higher depression
* Unable to read, write, and speak in English
* Unable to provide consent
* Do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of depression | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in symptoms of depression as measured by Beck Depression Inventory-FastScreen (7 items, possible range = 0-21)

SECONDARY OUTCOMES:
Change in symptoms of depression | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in symptoms of depression as measured by Patient Health Questionnaire-9 (9 items, range = 0-27)
Change in symptoms of depression, anxiety, and stress | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in symptoms of depression, anxiety, and stress as measured by Depression Anxiety Stress Scales-Short Form (21 items, range = 0-42 per depression, anxiety, or stress sub-scale)
Change in positive affect | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in positive affect, as measured by the Positive and Negative Affect Schedule, positive affect sub-scale (10 items, range = 10-50)
Change in negative affect | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in negative affect, as measured by the Positive and Negative Affect Schedule, negative affect sub-scale (10 items, range = 10-50)
Change in behavioral activation | Measured at baseline, 1-week, 2-week, 5-week. Outcome is change from baseline to each of the subsequent time points.
  Change in behavioral activation, as measured by the Behavioral Activation for Depression Scale - Short Form (9 items, range = 0-54)

OTHER OUTCOMES:
Intervention satisfaction | Measured at post-intervention (2-weeks)
  Satisfaction with the intervention, as measured with the mHealth Satisfaction Questionnaire (14 items, range = 14-70)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable request.

REFERENCES:
- Available data/document: Statistical Analysis Plan — https://osf.io/zw5cq